CLINICAL TRIAL: NCT01256073
Title: An Open-label, Safety and Tolerability Extension Trial Assessing Repeated Dosing of Anti-KIR (1-7F9) Human Monoclonal Antibody in Patients With Acute Myeloid Leukaemia
Brief Title: A Safety and Tolerability Extension Trial Assessing Repeated Dosing of Anti-KIR (1-7F9) Human Monoclonal Antibody in Patients With Acute Myeloid Leukaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH 2101-102
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — IPH-2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPH2101 (Experimental)
  Interventions: Drug: IPH2101

INTERVENTIONS:
Drug: IPH2101 — IPH2101 fully human anti-KIR monoclonal antibody

SUMMARY:
The trial is a multi-centre, open-label, safety and tolerability extension trial to the IPH2101-101 (previously NN1975-1733) first human dose trial completed with a larger subject pool at an optimal dose level. The trial is conducted in elderly Acute Myeloid Leukemia (AML) patients over the age of 60 years, in complete remission, and who are not eligible for allogeneic stem-cell transplantation. The dose given to the individual patient will be the same as the patient received in the single dose trial IPH2101-101 and 1 mg/kg or 2 mg/kg for the 12 patients in an additional cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
2. Acute myeloid leukaemia (AML) according to WHO Criteria
3. Morphological complete remission (CR) defined according to NCI criteria, or CRi with incomplete platelet count recovery only after 1 or 2 cycles of induction chemotherapy, and at least 1, and maximally 6 cycles of consolidation chemotherapy:

   * Absolute neutrophile count > 1x 109/L
   * Platelets > 80x109/L
   * Independency of blood transfusions
   * Less than 5% blasts in bone-marrow
   * No Auer rods
   * No symptoms of disease
4. Life expectancy > 4 months as judged by the Investigator
5. The patient is > or = 60 years of age but < or = 80 years of age
6. The patient has completed participation in the IPH2101-101(previously NN1975-1733)trial with an acceptable safety profile, as judged by the Investigator or is screened for the additional cohort
7. Time since last dose of chemotherapy at least 30 days and no more than 60 days if the patient did not participate in IPH2101-101 trial before
8. Recovery from acute toxicities of all previous anti-leukaemic therapies
9. KIR-expression on patient NK-cells (ability to bind Anti-KIR(1-7F9)) if the patient did not participate in IPH2101-101 trial before
10. ECOG performance status 0, 1 or 2
11. No major organ dysfunction as judged by the Investigator
12. The patients must have the following clinical laboratory values:

    * Serum creatinine < or = 2 md/dL
    * Total bilirubin < or = 1.5 x the upper limit of normal
    * Asparatate aminotransferase (AST) < 3x the upper limit of normal

Exclusion Criteria:

1. Known or suspected allergy to trial product or related products
2. Previous participation in this trial
3. AML classified as FAB M3 (APL, acute promyelocytic leukaemia) or with good prognosis AML i.e. t(8;21)(q22;q22) or inv(16)(p13q22) or t(16;16)(p13;q22) or their molecular equivalents
4. Eligibility for allogeneic haematopoietic transplantation
5. The patient is currently receiving, or has within the last 4 weeks received other investigational anti-leukemic treatment such as cytokine treatment, except Anti-KIR(1-7F9)
6. The patient has received G-CSF treatment within the last 30 days prior to screening
7. Systemic steroid treatment within the last 4 weeks prior to screening
8. Patient has active autoimmune disease
9. Diagnosis of monoclonal gammopathy
10. Patient has active infectious disease
11. Previous leukaemic CNS involvement
12. Cardiac failure (New York Heart Association [NYHA] grade III-IV)
13. Left ventricular ejection fraction (LVEF) less than 45 % of normal evaluated by ultrasound or isotopic evaluation
14. Severe neurological/psychiatric disorder
15. HIV or chronic hepatitis infection
16. Clinical evidence of an active second malignancy
17. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
18. Any new medical condition that in the opinion of the Investigator disqualifies the patient for inclusion

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of repeating dosings of Anti-KIR(1-7F9) | every 2 weeks
  using the US National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
To assess the pharmacokinetics upon repeated dosing(s)of Anti-KIR(1-7F9) | every 2 weeks
To assess the pharmacodynamics upon repeated dosing(s) of Anti-KIR(1-7F9) | every 2 or 4 weeks
  * Degree of KIR-occupancy on patient NK-cells
  * Plasma inflammatory cytokines (IFN-γ, TNF-α, IL-1, IL-6)
  * Immunophenotyping (NK-, B- and T-lymphocyte counts and activation status)
  * NK-cell surface markers (activation markers and inhibitory receptors)
  * Functional assay of NK-cell activity only for patient from additional cohort
To assess signs of efficacy of repeated dosing(s) with Anti-KIR(1-7F9) | to date of progression diagnosed or until death
  * Reduction in minimal residual disease measured by WT-1 expression in blood and bone marrow
  * Progression-free survival (measured as calendar days from the first dosing of Anti-KIR(1-7F9) (in the IPH2101-101 trial) to date of progression diagnosed or until death by any cause
  * Overall survival measured as calendar days from the first dosing of Anti-KIR (1-7F9) to date of death

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Vey, MD, Principal Investigator — Institut Paoli Calmettes Marseille France
Locations (6):
- France (6):
  - Institut Paoli-Calmettes, Marseille, Marseille Cedex 09
  - Hopital Dupuytren, Limoges
  - C.H.R.U. de Nantes - Hotel Dieu, Nantes
  - Centre Hospitalier Lyon Sud - Hospices Civils de Lyon, Pierre-Bénite
  - Hopital de Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif